CLINICAL TRIAL: NCT02413801
Title: Serum, Cellular and Imaging Markers of Arthritis in Psoriasis Patients
Acronym: RRF
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Rheumatology Research Foundation (Other)
Responsible Party: Principal Investigator, Christopher Ritchlin, M.D., M.P.H.; Professor of Medicine, Chief of Allergy, Immunology & Rheumatology Division, University of Rochester
Other Study IDs: RSRB 53131
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2024-06

CONDITIONS: Psoriasis
Keywords: Psoriasis; PDUS
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and bone marrow samples that remain after study assays are completed may be stored for future non-genetic research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Psoriasis: Individuals with psoriasis
- Healthy: Individuals that are healthy

SUMMARY:
The events that underlie the conversion from Psoriasis to Psoriatic Arthritis (PsA) are not well understood. This conversion occurs 30% of the time within the first 10 years of psoriasis diagnosis. PsA patients have about a 50% chance of developing joint damage within the first 2 years of disease. A biomarker that identifies subclinical joint inflammation in psoriasis patients would allow for a diagnostic tool to allow for earlier intervention in psoriasis patients and provide a better understanding of the underlying molecular pathogenesis that may lead to development of new therapeutic targets in PsA.

DETAILED DESCRIPTION:
Our long-term goals are to: 1) develop arthritis biomarkers in psoriasis patients that will facilitate early treatment interventions; and, 2) identify new therapeutic targets in PsA through better understanding of the underlying molecular pathogenesis. PsA, an inflammatory arthritis associated with psoriasis, affects approximately 650,000 adults in the United States and is associated with increased morbidity and mortality. Joint inflammation and damage arise within the first 2 years of disease in 50% of patients who manifest bone erosions and joint space narrowing on plain x-rays. The advent of Tumor Necrosis Factor antagonists (TNFi) for treatment of PsA has dramatically improved clinical response and slowed bone and cartilage degradation. Nevertheless, up to 45% of patients do not meet primary endpoints in clinical trials, which underscores the need for new therapeutic options.

Another approach to improve treatment response is early PsA diagnosis, and recent data indicate that treatment soon after disease onset can improve outcomes. Relevant to the potential for early intervention and prevention, psoriatic skin plaques typically precede PsA by 10 years. Moreover, a significant percentage of these psoriasis patients have subclinical musculoskeletal imaging findings. These findings provide an unparalleled opportunity for early intervention that could potentially limit or halt joint inflammation and damage. Regrettably, despite the obvious advantages of early diagnosis and treatment, this goal remains elusive because the clinical significance of imaging abnormalities in psoriasis remains unknown. Furthermore, investigators have limited understanding of the mechanisms that underlie the transition from psoriasis to PsA, and investigators lack the disease specific biomarkers necessary to identify psoriasis patients with new onset arthritis or sub-clinical disease. Lastly, up to a third of psoriasis patients with moderate to severe skin disease report they are undertreated and many are on topical agents unlikely to have a significant effect on subclinical or clinically apparent joint inflammation.

Up to 150 subjects will be consented and studied in this cross-sectional study - 125 subjects with Psoriasis (Ps) and 25 Healthy controls. Power Doppler Ultrasound (PDUS) in joints and entheses will be analyzed to find at least 35 subjects with positive US findings defined as synovitis, effusion, joint erosions, or increased vascularity otherwise known as a signal. Up to 50 Ps patients with positive PDUS results will be followed prospectively and contacted at intervals to update medication history indefinitely. Ps patients will be asked for a follow up PDUS 4 months post start of biologic, DMARD therapy or phototherapy if the patient decides to go on such therapies to study longitudinally.

Up to 30 bone marrow aspirations on healthy and PDUS positive Psoriasis subjects will be performed. A bone marrow aspiration post start of biologic or DMARD standard of care therapy will be assessed as well.

Research assays: serum will be used to measure biomarker 14-3-3η levels, which may be analyzed by an external company. Peripheral blood will be used to measure the frequency of DC-STAMP+ cells (CD14+DC-STAMP+ CD4+DCSTAMP+DC-STAMP+IL-17+). Using multichromatic flow cytometry, we will measure DC-STAMP expression on peripheral blood cells and on bone marrow cells. To determine if elevated BM DC-STAMP expression by stromal cells, T cells and/or monocytes promotes OC formation, co-cultures of bone marrow stromal and hematopoietic cells with peripheral blood cells will be analyzed for OCPs.

ELIGIBILITY:
Inclusion Criteria:

* All Subjects

  1. Ability to provide written informed consent
  2. Subjects must be 18 years old or older
* Psoriasis Subjects

  1. Patients with self-diagnosed Psoriasis. These subjects may present with thick, scaly, silvery and/or red skin, without ever having been diagnosed by a dermatologist:

     * Starting either a DMARD or biologic standard of care for their psoriasis OR
     * Currently started taking a DMARD within the last two weeks of study visit procedures OR
     * Currently not using a DMARD or biologic treatment, subjects may be using topical creams or UV therapy
  2. Willing to be studied longitudinally with a 4 month follow-up blood draw and PDUS if initial PDUS demonstrates positive findings.
* Bone Marrow Aspiration:

  1. Willing to undergo procedure.
  2. Psoriasis: positive findings on Power Doppler Ultra Sound (PDUS+) such as joint erosion, effusion, synovitis or increased vascularity, otherwise known as a signal.

Exclusion Criteria:

* All Subjects

  1. Unable to donate blood because of poor venous access or intolerance of phlebotomy.
  2. Chronic pain syndrome, autoimmune or active inflammatory conditions other than the conditions being studied. (i.e., chronic infection with hepatitis B or hepatitis C, inflammatory arthritis, etc) which in the investigator's opinion may confound the study results.
* Healthy subjects:

  1. Musculoskeletal conditions such as joint pains or swelling, fracture, tendonitis or trauma in the past 3 months, gout, or any arthritis which in the investigator's opinion may confound the study results.
  2. Illness in the last month which in the investigator's opinion may confound the study results.
  3. Taking systemic steroids or immunosuppressants
* Psoriasis Subjects:

  1. Evidence of inflammatory arthritis.
  2. Psoriatic Arthritis Screening and Evaluation (PASE) questionnaire score greater than or equal to 47.
  3. Meet CASPAR criteria for PsA.
* Bone Marrow Aspiration:

  1. Side effect to local anesthetics such as lidocaine or novocain.
  2. Bleeding disorders or conditions requiring treatment with, NSAID, aspirin, anti-coagulants or anti-platelet agent, unless a physician investigator determines it to be safe to hold these agents for 2 weeks.
  3. Known thrombocytopenia (< 100,000) or clinically significant PT or PTT outside the normal range.
  4. Pregnant women should not participate; Pregnancy tests will not be performed.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female subjects that are 18 years old and older. Due to the demographic distribution of the disease we expect all or nearly all subjects to be Caucasian, however no subjects will be excluded from any group based on race or ethnic origin.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Correlation of abnormal ultrasound signals with peripheral blood in subclinical PsA | Week 0
  To examine if subclinical PsA, as measured by abnormal ultrasound signals, correlate with peripheral blood cellular and serologic biomarkers of inflammation and joint damage. Power Doppler Ultrasound (PDUS) signals in joints and entheses of approximately 125 Ps pts in order to identify at least 35 pts with subclinical PsA (and 25 healthy controls). Investigators will compare both the frequency of DC-STAMP+ cells (CD14+DCSTAMP+ CD4+DC-STAMP+ DC-STAMP+IL-17+) and serum biomarker 14-3-3η levels between the Ps pts with subclinical PsA (PDUS+), up to 50 Ps pts without evidence of subclinical PsA (PDUS-), and controls.
To understand if systemic therapies for Ps can reduce subclinical joint inflammation. | Week 0 to week 16
  Investigators will monitor the change in PDUS signals and PB biomarkers in at least 35 subclinical PsA pts identified from baseline to month 4 following Phototherapy, DMARD or Biologic therapy.
To examine if DC-STAMP expression on BM cells is associated with subclinical PsA and increased OC formation in psoriasis. | Week 0 to week 16
  Investigators will analyze PB and BM DC-STAMP expression in PDUS+ pts evaluated at baseline and at 4 months post standard of care treatment. Then, to determine if elevated BM DC-STAMP expression by stromal cells, T cells and/or monocytes promotes OC formation, co-cultures of BM stromal and hematopoietic cells with PB cells will be analyzed for OCPs.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ritchlin, MD/MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Information of any type may be shared with researchers at other institutions. Subjects will be made aware of this in the informed consent form.
Time Frame: Once a subject signs the consent form to allow for sharing, any sample collected may be shared with collaborating institutions. This will last indefinitely or until the subject cancels consent to share.
Access Criteria: Only investigators that the study team collaborates with will have access to samples. Data will not include any information that is identifying.